CLINICAL TRIAL: NCT05555901
Title: The Efficacy and Safety of Fruquintinib Combined With Chemotherapy vs Bevacizumab Combined With Chemotherapy as Second-line Treatment in Patients With Metastatic Colorectal Cancer: A Prospective, Multi-center, Randomized Study
Brief Title: The Efficacy and Safety of Fruquintinib Plus Chemotherapy as Second-line Treatment in Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Deputy director of the department of general surgery, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FRESCO-3
Record Dates: First submitted 2022-09-22; First posted 2022-09-27 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Fruquintinib plus Chemotherapy; second-line treatment
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: fruquintinib plus chemotherapy vs bevacizumab plus chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fruquintinib+ chemotherapy (Experimental): Patients will receive fruquintinib+ FOLFIRI once every four weeks as the second-line treatment. After receiving 4-6 months of second-line treatment, patients who achieve disease control will receive fruquintinib + capecitabine as maintenance treatment.
  Interventions: Drug: Fruquintinib+ chemotherapy
- Bevacizumab+ chemotherapy (Active Comparator): Patients will receive bevacizumab+ FOLFIRI once every two weeks as the second-line treatment. After receiving 4-6 months of second-line treatment, patients who achieve disease control will receive bevacizumab + capecitabine as maintenance treatment.
  Interventions: Drug: Bevacizumab+ chemotherapy

INTERVENTIONS:
Drug: Fruquintinib+ chemotherapy — Second-line treatment : Fruquintinib+FOLFIRI Drug: Fruquintinib 4mg, orally, once daily, 3 weeks on/ 1 week off, q4w
  Drug: FOLFIRI regimen Irinotecan 180 mg/m2, and LV 400 mg/m2 followed by bolus 5-fluorouracil 400mg/m2 and a 46-48-hour continuous infusion 2400mg/m2 5-fluorouracil on day 1, q2w
  Maintenance treatment：Fruquintinib+Capecitabine Drug: Fruquintinib 4mg, orally, once daily, 2 weeks on/ 1 week off, q3w Drug: Capecitabine 825 mg/m2, orally, twice daily, q3w
  Arms: Fruquintinib+ chemotherapy
Drug: Bevacizumab+ chemotherapy — Second-line treatment : Bevacizumab+FOLFIRI Drug: Bevacizumab 5mg/kg on day 1, q2w
  Drug: FOLFIRI regimen Irinotecan 180 mg/m2, and LV 400 mg/m2 followed by bolus 5-fluorouracil 400mg/m2 and a 46-48-hour continuous infusion 2400mg/m2 5-fluorouracil on day 1, q2w
  Maintenance treatment：Bevacizumab+Capecitabine Drug: Bevacizumab 7.5mg/kg on day 1, q3w Drug: Capecitabine 825 mg/m2, orally, twice daily, q3w
  Arms: Bevacizumab+ chemotherapy

SUMMARY:
This is a prospective, multi-center, randomized study evaluating the efficacy and safety of fruquintinib combined with chemotherapy vs bevacizumab combined with chemotherapy as second-line treatment in patients with metastatic colorectal cancer. Patients will receive fruquintinib+ FOLFIRI or bevacizumab+FOLFIRI as the second-line treatment. After receiving 4-6 months of second-line treatment, patients who achieve disease control will receive fruquintinib + capecitabine or bevacizumab+ capecitabine as maintenance treatment. All patients will be treated until progressive disease, death from any cause, unacceptable toxicity or informed consent withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-75years (inclusive);
* Body weight ≥40 kg;
* Histological or cytological confirmed colorectal cancer;
* Expected survival >12 weeks;
* Fail in previous first-line standard therapy, which must include a fluorouracil (5-fluorouracil or capecitabine), oxaliplatin ;
* At least one measurable lesion (according to RECIST1.1);
* Adequate hepatic, renal, heart, and hematologic functions;
* Negative serum pregnancy test at screening for women of childbearing potential.

Exclusion Criteria:

* Received radiation therapy, surgical procedure, chemotherapy, immunotherapy or molecular targeted therapy, or other investigational drugs within 4 weeks prior to treatment
* Prior treatment with anti-angiogenic small molecule targeted drugs, such as fruquintinib, etc
* Prior treatment with an irinotecan-based chemotherapy regimen
* Symptomatic brain or meningeal metastases (except for patients with BMS who have received local radiotherapy or surgery for more than 6 months and whose disease is stable);
* Patients with hypertension that cannot be well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg)
* Have obvious clinical bleeding symptoms or obvious bleeding tendency within 3 months before treatment (bleeding > 30 mL within 3 months, hematemesis, black feces, hematozoia), hemoptysis (fresh blood > 5 mL within 4 weeks), etc. Treatment for venous/venous thrombosis events within the previous 6 months, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism; Long-term anticoagulant therapy with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day);
* Tumor invasion of large vascular structures, such as pulmonary artery, superior vena cava or inferior vena cava, was found during screening, which was judged by the investigator to have a greater risk of bleeding;
* Active heart disease, including myocardial infarction, severe/unstable angina, 6 months prior to treatment. Echocardiography examination left ventricular ejection fraction < 50%, arrhythmia control is not good;
* The patient has had other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix);
* Allergy to the study drug or any of its excipients;
* Severe infection with active or uncontrolled infection;
* Any other disease, with clinical significance of metabolic abnormalities, abnormal physical examination or laboratory abnormalities, according to researchers, there is reason to suspect the patient has not suitable for the use of study drugs of a disease or condition (such as have a seizure and require treatment), or will affect the interpretation of results, or to make patients in high-risk situations;
* Urine routine showed urine protein ≥2+, and 24-hour urine protein level >1.0g.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2023-06-18 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  time from randomization to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

SECONDARY OUTCOMES:
Objective response rate (ORR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  the proportion of patients with complete response or partial response, using RECIST v 1.1.
Disease Control Rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 1 year
  the proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1.
Overall survival (OS) | from randomization until death due to any cause, assessed up to 2 year
  time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Locations (13):
- China (13):
  - The First Hospital of Putian City, Putian, Fujian
  - The Fourth Hospital of Hebei Medical University and Hebei Tumor Hospital, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Qilu Hospital of Shandong University (QLH), Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Renji hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Changhai Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital Affiliated to The Shanghai Jiao Tong University Medical School, Shanghai, Shanghai Municipality
  - the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - Zhongshan hosptial, Fudan University, Shanghai